CLINICAL TRIAL: NCT03246139
Title: Action Observation, Imagery and Execution as a New Intervention Strategy for Stroke Rehabilitation: Short- and Long-term Treatment Effects and Neural Mechanism
Brief Title: Action Observation, Imagery and Execution for Stroke Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201602056A3; N201705016 (Other: Taipei Medical University - JointInstitutional Review Board)
Record Dates: First submitted 2017-08-03; First posted 2017-08-11 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-06

CONDITIONS: Stroke
Keywords: stroke; neurorehabilitation; mirror neuron system; action observation; motor imagery; MEG
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Action observation, imagery & execution (Experimental)
  Interventions: Behavioral: Action observation, imagery & execution
- Action observation (Active Comparator)
  Interventions: Behavioral: Action observation
- Control treatment (Active Comparator)
  Interventions: Behavioral: Control treatment

INTERVENTIONS:
Behavioral: Action observation, imagery & execution — The participants will be asked to observe movements through a video clip, practice motor imagery, and executing the movements that the participants observed.
  Arms: Action observation, imagery & execution
Behavioral: Action observation — The participants will be asked to observe videos and then practice what the participants observed.
  Arms: Action observation
Behavioral: Control treatment — The participants will receive UE training without watching videos or imagining movements/tasks.
  Arms: Control treatment

SUMMARY:
The specific study aims will be:

1. To investigate the short- and long-term treatment effects of action observation, imagery, and execution therapy (AOIE) compared with an action observation therapy (AO) group and a control treatment group as controls on different aspects of outcomes in patients with stroke.
2. To examine the neural mechanisms and changes in cortical neural activity after the interventions in stroke patients.
3. To examine the correlations between AOIE-induced brain activation changes and the clinical efficacy of AOIE.
4. To identify who are the possible good responders to the therapy based on baseline motor function and motor imagery ability of the participants.

DETAILED DESCRIPTION:
The investigators propose a 3-year randomized controlled trial to (1) investigate the short- and long-term treatment efficacy of AOIE, action observation alone, versus control treatment on clinical outcomes of patients with subacute stroke, (2) examine the neural mechanisms and activation changes after the 3 interventions by using an advanced brain imaging technique, magnetoencephalography (MEG), (3) determine the correlations between neural activation changes and clinical outcomes, and (4) identify who are the good responders to the AOIE therapy. An estimated total of 96 patients with subacute stroke will be recruited in this study. All participants will be randomly assigned to receive 1 of the 3 interventions for 3 weeks (a total of 15 sessions). Clinical outcome measures will be conducted at baseline, immediately after treatment (3 weeks), and at 3 months follow-up. The MEG assessment will be conducted at baseline and immediately after treatment (3 weeks). For the MEG study, The investigators anticipate to enroll 12 to 15 patients in each group to complete neuroimaging evaluation because of the specific eligibility criteria and high costs of MEG. The patients can still participate in the study, receiving rehabilitation therapy and clinical evaluations, even if the participants will not be included in the MEG study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as having a unilateral stroke;
* 1 to 12 months after stroke onset
* from 20 to 80 years of age
* a baseline score of the Fugl-Meyer Assessment (FMA) of 20 to 60
* able to follow the study instructions
* capable of participating in therapy and assessment sessions.

Exclusion Criteria:

* patients with global or receptive aphasia,
* severe neglect
* major medical problems, or comorbidities that influenced UE usage or caused severe pain

Additionally, if patients have no metal implants, no head traumas or neurosurgical operations, and can perform MEG motor tasks, the participants can additionally participate in the MEG assessment.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change scores of Modified Rankin Scale | baseline, 3 weeks , 3 months
  The Modified Rankin Scale is used to assess the degree of stroke disability.
Change scores of Fugl-Meyer Assessment | baseline, 3 weeks , 3 months
  Change from baseline motor impairment at 3 weeks on the Fugl-Meyer Assessment.

SECONDARY OUTCOMES:
Change scores of Box and Block Test | baseline, 3 weeks , 3 months
  The Box and Block Test is a measure of hand dexterity with satisfactory reliability and validity in patients with stroke.
Change scores of Chedoke Arm and Hand Activity Inventory (CAHAI) | baseline, 3 weeks , 3 months
  The CAHAI measures the upper-limb motor function after stroke.
Change scores of Movement Imagery Questionnaire, revised second version | baseline, 3 weeks , 3 months
  The MIQ-RS will be applied to assess patient's ability of motor imagery.
Change scores of Functional Independence Measure | baseline, 3 weeks , 3 months
  The Functional Independence Measure is a frequently used scale to assess basic activities of daily function.
Change scores of physical intensity measured by activity monitors | baseline, 3 weeks , 3 months
  The accelerometers (ActiGraph) are used to provide an objective measure of the amount of the affected arm in patient's real-life environments. The parameter of average intensity of physical activity (counts/minute) will be reported.
Change scores of energy expenditure measured by activity monitors | baseline, 3 weeks , 3 months
  The accelerometers (ActiGraph) are used to provide an objective measure of the amount of the affected arm in patient's real-life environments. The parameter of energy expenditure(Kcal) will be reported.
Change scores of Stroke Impact Scale (SIS) Version 3.0 | baseline, 3 weeks , 3 months
  The Stroke Impact Scale Version 3.0 is a patient-reported outcome to evaluate function, participation, and health-related quality of life of stroke survivors with sound psychometric properties.
Magnetoencephalography (MEG) | baseline, 3 weeks
  Magnetoencephalography (MEG) can directly measure cortical neural activity and detect the oscillatory signals mainly by the changes in the postsynaptic fields of pyramidal cells. The MEG assessment will be conducted at baseline and immediately after treatment (3 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Wei Hsieh, PhD, Principal Investigator — Department of Occupational Therapy and Graduate Institute of Behavioral Sciences, College of Medicine, and Healthy Aging Research Center, Chang Gung University
Locations (4):
- Taiwan (4):
  - Taipei medical university hospital, Taipei
  - Taipei Medical University Shuang Ho Hospital, Taipei
  - Taoyuan Chang Gung Memorial Hospital, Taoyuan
  - Lo-Sheng Sanatorium and Hospital, Ministry of Health and Welfare, Taoyuan

IPD SHARING:
Plan to Share IPD: No